CLINICAL TRIAL: NCT01464853
Title: Effect of Enteral Nutrition Support for Critically Ill Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis indicated significant additional subjects needed to demonsate statistical difference in primary outcome.
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK54
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-03

CONDITIONS: Respiratory Distress Syndrome,Adult; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Enteral Nutrition; Fatty Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specialized Enteral Nutrition (Experimental): Enteral Feeding to provide 25 kcal/Kg/day
  Interventions: Other: Enteral nutrition with fatty acids
- Standard Enteral Nutrition (Active Comparator): Enteral Feeding to provide 25 kcal/Kg/day
  Interventions: Other: Standard Enteral Nutrition

INTERVENTIONS:
Other: Enteral nutrition with fatty acids — Enteral Feeding to provide 25 kcal/Kg/day
  Arms: Specialized Enteral Nutrition
Other: Standard Enteral Nutrition — Enteral Feeding to provide 25 kcal/Kg/day
  Arms: Standard Enteral Nutrition

SUMMARY:
To determine whether specialized enteral nutrition support can improve oxygenation status in critically ill patients with acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) comparing to a standard enteral nutritional formula.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female.
2. ALI or ARDS
3. PaO2/FiO2 > 100 and ≤ 300 torr.
4. Evidence of bilateral pulmonary infiltrates/opacity on chest radiograph.
5. Enteral access
6. Systemic inflammatory response syndrome (SIRS) - two or more of the following must be present:

   1. Body temperature less than 36°C or greater than 38°C
   2. Heart rate > 90 beats per minute
   3. Tachypnea with > 20 breaths per minute; or an arterial partial pressure of carbon dioxide < 4.3 kPa (32 mmHg)
   4. White blood cell count < 4000 cells/mm³ or > 12,000 cells/mm³; or the presence of > 10% immature neutrophils.

Exclusion Criteria:

1. Dialysis for renal failure
2. Unable to initiate Enteral feeding within 48 hours since all inclusion criteria met.
3. Anticipated life expectancy less than 24 hours.
4. Patient with severe chronic liver disease
5. Neuromuscular disease that impairs ability to ventilate without assistance
6. Head trauma and/or drowning with a Glasgow coma score of 5
7. Receiving intravenous lipid emulsions from parenteral nutrition within 12 hours of baseline.
8. Receiving propofol
9. Airway reconstructive surgery.
10. Malignancy or irreversible disease for which 6-month mortality is greater than 50%.
11. Burns greater than 25% total body surface area.
12. Unwillingness or inability to utilize the ARDS network ventilation protocol.
13. HIV positive.
14. Chronic mechanical ventilation.
15. Severe, acute pancreatitis.
16. Refractory shock
17. Congestive heart failure with pulmonary edema as the primary cause of hypoxemia.
18. Acute myocardial infarction or cardiac surgery within 7 days.
19. Solid organ transplant.
20. INR > 5.0 or platelet count < 30,000/mm3 or history of bleeding disorder.
21. Intracranial hemorrhage within the past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Oxygenation status improvement | 28 days

SECONDARY OUTCOMES:
Length of ventilation | 28 days
Length of ICU stay | 28 days
Incidence of organ failures | 28 days
Incidence of ventilator-associated pneumonia | 28 days
Mortality | 28 days
Glycemic control | 28 days
Inflammation | 28 days
Vitamin D status | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Luo, MD, PhD, Study Chair — Abbott Nutrition
Locations (9):
- Russia (9):
  - 1st City Clinical Emergency Hospital n.a. E.E. Volosevich, Arkhangelsk
  - City Clinical Hospital #2, Krasnodar
  - Krasnoyarsk State Medical University n.a. Prof V.F. Voyno-Yasenetskogo, Krasnoyarsk
  - Central Clinical Hospital #1, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Clinical Medical Unit #1, Perm
  - St. Petersburg Scientific Research Institute of Emergency Care n.a. I.I.Dzhanelidze, Saint Petersburg
  - Republican Clinical Hospital n.a. G.G. Kuvatova, Ufa
  - Central City Hospital #7, Yekaterinburg